CLINICAL TRIAL: NCT00556751
Title: Epidemiology and Mechanisms of ECG Abnormalities: Young Adulthood to Middle Age
Brief Title: Evaluating Electrocardiogram (ECG) Abnormalities From Young Adulthood Through Middle Age
Acronym: CARDIA ECG
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1406; R01HL086792 (NIH)
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2007-12

CONDITIONS: Cardiovascular Diseases
Keywords: Electrocardiogram; Electrocardiography; Cardiovascular Risk Factors; Cholesterol; Blood Pressure; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An electrocardiogram (ECG) is a test that evaluates the electrical activity of the heart and can be used to detect heart problems. By analyzing ECGs collected over a 20-year period, this study will examine ECG abnormalities and the differences in ECG findings between black and white people, from young adulthood through middle age.

DETAILED DESCRIPTION:
An ECG is a test that detects and records the electrical activity of the heart. As a diagnostic tool, it can detect and locate the source of heart problems, including heart attacks, irregular heart beats, cardiovascular disease, or other abnormalities of the heart. An ECG procedure involves attaching electrodes to the skin on the chest, arms, and legs while the electrodes detect electrical signals of the heart, and a machine displays the signals on a computer screen and graph paper. An ECG may be a beneficial way to detect cardiovascular disease because it is a low-cost and non-invasive test that is widely available in the clinical setting.

This study will examine ECGs and other study data from participants in the Coronary Artery Risk Development in Young Adults (CARDIA) study. As ECG abnormalities typically begin to develop in young adults, the CARDIA participants will provide researchers with an excellent study population. As part of the CARDIA study, ECGs were obtained from participants at baseline, and Years 7 and 20. Study researchers will use state-of-the-art technology and standardized Minnesota Code and Novacode methods to electronically code participants' ECGs and accomplish the following: 1) assess the frequency of ECG abnormalities in young adults of different races; 2) examine potential risk factors for the development and progression of ECG abnormalities; 3) investigate the relationship between ECG abnormalities and other measures of heart disease; and 4) assess differences in the frequency and patterns of ECG abnormalities between different racial groups. Study researchers will also analyze additional CARDIA study data, including cardiovascular disease risk factors, measures of atherosclerosis, and echocardiographic ultrasound pictures of the heart.

This research will provide important insights into the ways in which ECG abnormalities are associated with increased risk for cardiovascular disease and how the risk may differ between blacks and whites. Results from this study may ultimately lead to improvements in preventive strategies for cardiovascular disease in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the CARDIA study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CARDIA study participants, which included black and white men and women, 18- to 30-years-old at the time of study entry from 1985 to 1986, and balanced on sex, race, and education status
Sampling Method: Non-Probability Sample
Enrollment: 5115 (Actual)
Dates: Start 1985-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Development of resting ECG abnormalities, specifically isolated non-specific ST-segment and T-wave abnormalities | Measured at Years 7 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Donald M. Lloyd-Jones, MD, ScM, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Cutter GR, Burke GL, Dyer AR, Friedman GD, Hilner JE, Hughes GH, Hulley SB, Jacobs DR Jr, Liu K, Manolio TA, et al. Cardiovascular risk factors in young adults. The CARDIA baseline monograph. Control Clin Trials. 1991 Feb;12(1 Suppl):1S-77S. doi: 10.1016/0197-2456(91)90002-4. No abstract available. PMID 1851696